CLINICAL TRIAL: NCT07300501
Title: Stereotactic Aspiration of Brain Stem Hematoma: a Prospective, Multi-center, Randomized Controlled Trial
Brief Title: Stereotactic Aspiration of Brain Stem Hematoma
Acronym: SABSH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: RenJi Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Taizhou First People's Hospital (Other); Shenzhen Second People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Henan Provincial People's Hospital (Other); Zhujiang Hospital (Other); Xiangya Hospital of Central South University (Other); Qilu Hospital of Shandong University (Other); Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT20250094C-R1-3.0
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-08

CONDITIONS: Brain Stem Hematoma
Keywords: brain stem hematoma; Stereotactic aspiration; randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Treatment Group (No Intervention): The Conservative Treatment Group will adhere to the guideline-recommended standard management protocol for intracerebral hemorrhage.
- Stereotactic Aspiration Group (Experimental): In addition to receiving the guideline-recommended management for intracerebral hemorrhage, patients in the Stereotactic Aspiration Group will undergo stereotactic aspiration surgery as a routine intervention.
  Interventions: Procedure: stereotactic aspiration surgery

INTERVENTIONS:
Procedure: stereotactic aspiration surgery — Stereotactic aspiration of the brainstem hematoma is performed with the aid of a surgical robot for precise localization.
  Arms: Stereotactic Aspiration Group

SUMMARY:
This clinical study is a high-level evidence-based medical research project designed to compare the efficacy differences between stereotactic aspiration and conservative treatment in patients with brainstem hemorrhage. Brainstem hemorrhage is a life-threatening condition with extremely high rates of mortality and disability. Currently, there is ongoing debate regarding its treatment strategies, particularly the necessity of surgical intervention. Although surgical explorations have been conducted in China, there is a lack of high-quality, multi-center randomized controlled trial (RCT) evidence.

To address this, the present study was initiated by the First Affiliated Hospital, Zhejiang University School of Medicine, in collaboration with dozens of leading medical centers across China. The study adopts a prospective, multi-center, single-blind, randomized controlled design. It plans to enroll 300 eligible patients with primary brainstem hemorrhage, who will be randomly assigned to either the stereotactic aspiration treatment group or the conservative treatment group.

Key inclusion criteria are: radiologically confirmed brainstem hematoma volume >5 ml; hospital admission within 24 hours of onset; Glasgow Coma Scale (GCS) score of 4-8; National Institutes of Health Stroke Scale (NIHSS) score ≥21; age between 18 and 65 years; and presence of spontaneous respiration.

The primary endpoint of the study is the Modified Rankin Scale (MRS) score at 3 months post-treatment, which assesses neurological recovery and the degree of disability. Secondary endpoints include the incidence of complications such as acute hydrocephalus, intracranial infection, pulmonary infection, and re-bleeding, as well as the length of ICU stay and total hospital stay.

The study will strictly implement randomization and blinding procedures. Randomization will be centrally managed by the principal center, and outcome assessors will be blinded to ensure the objectivity and scientific rigor of the data. All participating centers are required to have extensive experience in minimally invasive treatment of brainstem hemorrhage. The study is expected to last for 3 years, encompassing phases for patient recruitment, treatment implementation, data collection, and statistical analysis.

The findings of this study are expected to provide high-level evidence-based medical evidence for the challenging clinical problem of brainstem hemorrhage, clarify the therapeutic value of stereotactic minimally invasive surgery, and thereby guide clinical practice and improve patient outcomes.

DETAILED DESCRIPTION:
1. Research Background and Rationale Primary brainstem hemorrhage (PBSH) represents the most severe and life-threatening form of spontaneous intracerebral hemorrhage. Due to its critical anatomical location involving vital centers, it is associated with high mortality (30-day mortality rates ranging from 47% to 80%) and extremely poor neurological outcomes. For a long time, the optimal treatment strategy for PBSH, particularly the value of surgical intervention, has been a subject of significant global controversy. Influential international guidelines, such as those from the American Heart Association/American Stroke Association (AHA/ASA), still regard surgery for PBSH as a relative or absolute contraindication, primarily due to the lack of high-level evidence.

   Concurrently, with advancements in neuroimaging, neuronavigation, and minimally invasive surgical techniques, several medical centers in China have progressively explored surgical interventions for PBSH, including stereotactic aspiration and neuroendoscopic evacuation, accumulating considerable clinical experience. The 2022 Chinese Expert Consensus on the Diagnosis and Treatment of Primary Brainstem Hemorrhage suggests that surgical treatment can be considered for specific patients, such as those with hematoma volume ≥5 ml and a Glasgow Coma Scale (GCS) score ≤7, following thorough assessment. However, the consensus is largely based on retrospective analyses or small case series, providing limited evidence that falls short of guiding widespread clinical practice.

   The core dilemma in current clinical decision-making lies in the disconnect between theory and practice. Theoretically, early hematoma evacuation may relieve compression on brainstem structures and facilitate neurological recovery. In practice, however, the risks inherent to surgery, heterogeneity in patient selection, variations in surgical timing and technique, and other factors leave it unclear whether surgical intervention offers a net clinical benefit. Therefore, conducting a rigorously designed and properly executed multicenter randomized controlled trial (RCT) to compare the impact of stereotactic minimally invasive aspiration versus standard medical conservative treatment on patient outcomes is of urgent and paramount importance. Such a study is essential to fill the existing evidence gap and establish a scientific treatment protocol.
2. Research Objectives and Core Content 2.1 Research Objective The primary objective of this study is to systematically compare the efficacy and safety of stereotactic brainstem hematoma aspiration versus conservative treatment alone in eligible patients with PBSH through a prospective, multicenter, randomized controlled trial. The focus is on evaluating the difference in the rate of death and disability (using the Modified Rankin Scale [MRS] score as the core metric) at 3 months post-treatment. The aim is to provide high-quality, generalizable evidence-based medical data to inform clinical decision-making for brainstem hemorrhage.

   2.2 Research Content

   This study focuses on the most challenging patient population in clinical practice: those with moderate-to-severe primary PBSH. By randomly assigning patients who meet strict inclusion and exclusion criteria to either the surgical intervention group (stereotactic aspiration) or the medical treatment group (standard conservative therapy), the study will objectively evaluate, within a unified and standardized treatment and follow-up framework:
   1. Whether surgical intervention can significantly improve patients' neurological functional outcomes (primary endpoint).
   2. Differences between the two groups in the incidence of various complications (e.g., re-bleeding, infection, hydrocephalus), length of intensive care unit (ICU) stay, and total hospital length of stay (secondary endpoints).
   3. The safety profile and spectrum of adverse events associated with surgical treatment.
3. Study Design and Methodological Highlights 3.1 Overall Design This is a multicenter, prospective, single-blind (with outcome assessors blinded), randomized controlled study.

   3.2 Subject Selection Inclusion Criteria: Precisely targets a population likely to benefit from intervention with relatively controllable risks. Criteria include: ① Primary PBSH confirmed by CT/MRI, with hematoma volume >5 ml; ② Time from onset to hospital admission and diagnosis within 24 hours; ③ Glasgow Coma Scale (GCS) score of 4-8 (moderate to severe coma); ④ National Institutes of Health Stroke Scale (NIHSS) score ≥21 (severe neurological deficit); ⑤ Age between 18 and 65 years; ⑥ Presence of spontaneous respiration upon admission.

   Exclusion Criteria: Aims to exclude cases of non-hypertensive hemorrhage, patients at high surgical risk, and those unable to complete follow-up. Criteria include: Hemorrhage caused by vascular malformation, cavernoma, or tumor stroke; presence of severe comorbidities such as significant cardiac, hepatic, or renal insufficiency, or malignant tumors; recent history of antiplatelet or anticoagulant medication use; and any condition expected to prevent completion of the 3-month follow-up.

   3.3 Randomization and Blinding Randomization: A central randomization system managed uniformly by the principal center (The First Affiliated Hospital, Zhejiang University School of Medicine) will be employed. Stratified randomization will be used, with age (18-45 years, 46-65 years) as the stratification factor to ensure baseline balance between the two groups. Participating centers will obtain treatment allocation results through this system upon patient enrollment.

   Blinding: A single-blind design will be implemented. The treating clinicians and the patients themselves will be aware of the group assignment (for ethical and practical reasons). However, the clinical research coordinators or assessors responsible for collecting data for the primary endpoint (MRS score) and some secondary endpoints will be blinded to group allocation to minimize assessment bias.

   3.4 Interventions Stereotactic Aspiration Group: In addition to standard medical treatment, this group will undergo "robot-assisted stereotactic brainstem hematoma aspiration + hematoma cavity drainage." The protocol emphasizes the use of stereotactic guidance systems to ensure surgical precision and safety.

   Conservative Treatment Group: This group will receive comprehensive, standardized medical management. The protocol details a full set of management measures, including blood pressure control, respiratory support, sedation and analgesia, hemostasis, stress ulcer prophylaxis, infection prevention, and venous thromboembolism prophylaxis.

   3.5 Endpoints Primary Endpoint: The Modified Rankin Scale (MRS) score at 3 months post-treatment. This internationally recognized scale is the core tool for assessing disability after stroke, scored from 0 to 6, with higher scores indicating greater disability or death. This study will analyze the distribution difference of MRS scores between the two groups.

   Secondary Endpoints: Encompass multiple dimensions of safety and healthcare resource utilization, including: ① Incidence of Complications: acute hydrocephalus, intracranial infection, pulmonary infection, re-bleeding; ② Hospitalization-related Metrics: length of ICU stay, total hospital length of stay; ③ Other physiological and laboratory parameters collected during hospitalization.

   3.6 Sample Size Calculation Based on preliminary trial data or previous literature and statistical analysis, the total sample size has been determined to be 300 patients, with 150 patients in each group.

   3.7 Study Flow and Follow-up
   1. Screening and Enrollment: Participating centers will conduct urgent screening of potentially eligible patients. Eligible patients who provide informed consent will be enrolled via the central randomization system.
   2. Treatment Phase: Patients will receive the assigned treatment according to the protocol and be closely monitored.
   3. Follow-up Phase: Key follow-up time points are established, including at enrollment (Day 0), Day 3, 1 month post-discharge (Day 30), and the primary endpoint assessment at 3 months (Day 90). MRS scores and other data will be collected through outpatient reviews or structured telephone follow-ups.
4. Data Management and Quality Control

   1. Data Collection: An Electronic Data Capture (EDC) system will be used with standardized Case Report Forms (CRFs).
   2. Quality Assurance: A detailed Quality Control Plan (QCP) will be developed and implemented. This includes routine remote data verification, periodic on-site monitoring, and potential data audits. All participating centers are required to be tertiary Grade A hospitals with experience in performing at least 10 minimally invasive procedures for PBSH annually to ensure technical homogeneity.
5. Ethical and Safety Considerations

   1. Ethical Review: The study protocol must be approved by the Institutional Review Board (IRB)/Ethics Committee of each participating center and filed with the clinical trial institution.
   2. Informed Consent: Written informed consent must be obtained from the patient or their legally authorized representative before any study-related procedures commence.
   3. Safety Monitoring: A strict system for reporting Adverse Events (AEs) and Serious Adverse Events (SAEs) will be established. All SAEs must be reported to the principal center and the local ethics committee within 24 hours. The protocol specifically outlines risks unique to brainstem puncture surgery (e.g., tract hemorrhage, brainstem injury) and corresponding management plans.
   4. Study Suspension/Termination Criteria: Clear criteria are defined for prematurely terminating the entire study due to safety concerns, administrative directives, or requests from ethics committees.
6. Research Team and Timeline

   1. Sponsor and Lead Center: The First Affiliated Hospital, Zhejiang University School of Medicine.
   2. Participating Centers: Dozens of leading neurosurgical centers across China, distributed in multiple regions, ensuring the study's representativeness and enrollment efficiency.
   3. Expected Timeline: The total study duration is planned for 3 years, specifically divided into: Preparation and Start-up Phase (6 months), Patient Recruitment and Treatment Phase (18 months), Data Cleaning and Analysis Phase (6 months), and Manuscript Writing and Publication Phase (6 months).
7. Expected Impact and Significance

This study is an ambitious and rigorously designed pivotal clinical trial initiated by the Chinese neurosurgical community targeting the "surgical no-go zone" of brainstem hemorrhage. Its anticipated outcomes are expected to have a significant impact in the following areas:

1. Providing High-Level Evidence: Generating the first multicenter RCT evidence on the efficacy of minimally invasive surgery for PBSH, directly challenging or validating current international and domestic guideline recommendations.
2. Guiding Clinical Practice: Clarifying the value of stereotactic aspiration in specific subgroups of PBSH patients, providing neurosurgeons and neurocritical care physicians with clear decision-making guidance.
3. Improving Patient Outcomes: If the study confirms a surgical benefit, it holds the potential to significantly reduce mortality and disability rates in these critically ill patients, alleviating the burden on families and society.
4. Promoting Technical Standardization: The standardized treatment protocols, surgical workflows, and perioperative management norms developed during the study can be promoted nationwide, elevating the overall diagnostic and therapeutic standards for this disease.

In conclusion, the successful implementation and completion of this study have the potential to resolve the therapeutic dilemma surrounding brainstem hemorrhage, representing an exploration of substantial clinical value and scientific significance.

ELIGIBILITY:
Inclusion Criteria:

* Primary PBSH confirmed by CT/MRI, with hematoma volume >5 ml;
* Time from onset to hospital admission and diagnosis within 24 hours;
* Glasgow Coma Scale (GCS) score of 4-8 (moderate to severe coma);
* National Institutes of Health Stroke Scale (NIHSS) score ≥21 (severe neurological deficit);
* Age between 18 and 65 years;
* Presence of spontaneous respiration upon admission.

Exclusion Criteria:

* Hemorrhage caused by vascular malformation, cavernoma, or tumor stroke;
* presence of severe comorbidities such as significant cardiac, hepatic, or renal insufficiency, or malignant tumors;
* recent history of antiplatelet or anticoagulant medication use;
* any condition expected to prevent completion of the 3-month follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Modified Rankin Scale (MRS) score at 3 months post-enrollment | at 3 months post-enrollment
  This internationally recognized scale is the core tool for assessing disability after stroke, scored from 0 to 6, with higher scores indicating greater disability or death. This study will analyze the distribution difference of MRS scores between the two groups.

SECONDARY OUTCOMES:
Incidence of complications | assessed at enrollment and again on the third day after enrollment
  Incidence of complications: acute hydrocephalus, intracranial infection, pulmonary infection, re-bleeding
Hospitalization-related Metrics | at 1 month and 3 months post-enrollment
  length of ICU stay, total hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng YANG, Doctor of Medicine, Principal Investigator — Zhejiang University
Locations (11):
- China (11):
  - The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Xiangya Hospital of Central South University, Changsha
  - Zhujiang Hospital,Southern Medical University, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Renji Hospital,School of Medicine,Shanghai Jiaotong University, Shanghai
  - Nanfang Hospital, Southern Medical University, Shenzhen
  - Shenzhen Second People's Hospital, Shenzhen
  - Taizhou First People's Hospital, Taizhou
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Xijing hospital, Xi'an
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymized Individual Participant Data (IPD) to promote scientific collaboration and transparency. The data sharing plan is as follows:
  1. What data will be shared? De-identified IPD underlying the results reported in the primary and secondary publications of this trial; The study protocol, statistical analysis plan , and informed consent form; The analytical code used to generate the results.
  2. When and how will data be available? Data will become accessible 12 months after the publication of the primary results of the trial. Requests can be submitted via email to the corresponding author or through a designated data repository platform.
  3. Additional protections:
  All shared data will be fully anonymized in accordance with applicable laws (China's Personal Information Protection Law) and international standards to protect participant privacy. Direct identifiers and any information with re-identification risk will be removed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become accessible 12 months after the publication of the primary results of the trial

REFERENCES:
- [Result] Wang SS, Yang Y, Velz J, Keller E, Luft AR, Regli L, Neidert MC, Bozinov O. Management of brainstem haemorrhages. Swiss Med Wkly. 2019 Apr 5;149:w20062. doi: 10.4414/smw.2019.20062. eCollection 2019 Mar 25. PMID 30950504
- [Result] Cavalcanti DD, Preul MC, Kalani MY, Spetzler RF. Microsurgical anatomy of safe entry zones to the brainstem. J Neurosurg. 2016 May;124(5):1359-76. doi: 10.3171/2015.4.JNS141945. Epub 2015 Oct 9. PMID 26452114
- [Result] Sun X, Zhu J, Lu M, Zhang Z, Li C, Zhan R. Robot-assisted puncture versus conservative treatment for severe brainstem hemorrhage: clinical outcomes comparison with experience of 138 cases in a single medical center. World J Emerg Surg. 2025 Feb 25;20(1):15. doi: 10.1186/s13017-025-00592-9. PMID 40001232
- [Result] Chen LH, Li FJ, Zhang HT, Chen WJ, Sun K, Xu RX. The microsurgical treatment for primary hypertensive brainstem hemorrhage: Experience with 52 patients. Asian J Surg. 2021 Jan;44(1):123-130. doi: 10.1016/j.asjsur.2020.04.016. Epub 2020 Jun 26. PMID 32600922
- [Result] Chen D, Tang Y, Nie H, Zhang P, Wang W, Dong Q, Wu G, Xue M, Tang Y, Liu W, Pan C, Tang Z. Primary Brainstem Hemorrhage: A Review of Prognostic Factors and Surgical Management. Front Neurol. 2021 Sep 10;12:727962. doi: 10.3389/fneur.2021.727962. eCollection 2021. PMID 34566872
- [Result] Li Y, Shang FJ, Xu Z, Wu DX, Li CH, Liu JF, Li YX, Zhang WH, Zhang WC. Comparison of stereotactic aspiration surgery and conventional treatment for primary brainstem haemorrhage. Clin Neurol Neurosurg. 2023 Nov;234:108008. doi: 10.1016/j.clineuro.2023.108008. Epub 2023 Oct 3. PMID 37866210